CLINICAL TRIAL: NCT05713370
Title: Sleep Restriction and Postprandial Lipemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2090503
Record Dates: First submitted 2023-01-13; First posted 2023-02-06 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Sleep Deprivation; Obesity
MeSH Terms: conditions — Sleep Deprivation; Obesity

STUDY DESIGN:
Intervention Model Description: Subjects will complete all arms of the study in a counterbalanced design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- no exercise, no SR (Placebo Comparator): 75 g of glucose will be given at the beginning of the study day (the evening prior there will be no exercise the night before the study day, normal sleep (8 h))
  Interventions: Dietary Supplement: high fat meal
- no exercise, SR (Experimental): 75 g of glucose will be given at the beginning of the study day (the evening prior there will be no exercise the night before the study day, 4 h of sleep the previous night)
  Interventions: Dietary Supplement: high fat meal
- Exercise, no SR (Experimental): 75 g of glucose will be given at the beginning of the study day (the evening prior there will be 45 min of exercise the night before the study day, normal sleep (8 h))
  Interventions: Dietary Supplement: high fat meal
- Exercise, SR (Experimental): 75 g of glucose will be given at the beginning of the study day (the evening prior there will be 45 min of exercise the night before the study day, 4 h of sleep the previous night)
  Interventions: Dietary Supplement: high fat meal

INTERVENTIONS:
Dietary Supplement: high fat meal — A high fat meal (milkshake) will be administered on the morning after the intervention of no exercise and no SR the night before.

SUMMARY:
Sleep restriction increases overnight and early morning non-esterified fatty acids (NEFA) levels, which are correlated with whole-body decreases in insulin sensitivity, consistent with the observed impairment of intracellular insulin signaling. Adipose tissue biopsies from sleep restricted subjects that are insulin stimulated have reduced phosphorylation of protein kinase B (pAKT). This protein is involved in suppression of intracellular lipolysis and NEFA release.

Aerobic exercise has beneficial effects on postprandial lipemia and insulinemia in normal-weight and obese individuals. Acute moderate-intensity aerobic exercise (30-90 min) performed 12-18 h before an oral fat tolerance test or mixed meal test reduces postprandial triglycerides (TG) and insulin concentrations. This response is largely dependent upon the exercise-induced energy deficit as the response is abolished when the calories expended during exercise are replaced.

However, it is not known if sleep restriction will interfere with the beneficial effects of prior exercise on postprandial lipemia. The aim of this project is to investigate if sleep restriction negates the positive effect that exercise has on postprandial lipemia. It is hypothesized that sleep restriction will negate the beneficial effects of prior exercise on postprandial lipemia. Additionally sleep restriction will result in a worsening of the lipid profile compared to no exercise.

For the proposed study, the investigators will use a repeated measures analysis of variance (ANOVA) (4 study conditions (no exercise+ sleep restriction, no exercise+normal sleep, exercise+normal sleep, exercise+sleep restriction) x time will be used to analyze changes in NEFA and TG concentrations while a one way ANOVA will be used to analyze area under the curve of the NEFA and TG concentrations.

DETAILED DESCRIPTION:
In the postprandial period, adipocytes respond to the increased insulin levels by suppressing intracellular triglycerides (TG) lipolysis and by increasing extracellular lipolysis by transporting lipoprotein lipase from intracellular vesicles to the surface of the endothelium. This results in decreased free fatty acids (FFA) release into the plasma and increased absorption of lipoprotein TGs, particularly those in chylomicrons and VLDLs.

Sleep restriction increases overnight and early morning non-esterified fatty acids (NEFA) levels, which are correlated with whole-body decreases in insulin sensitivity, consistent with the observed impairment of intracellular insulin signaling. Adipose tissue biopsies from sleep restricted subjects that are insulin stimulated have reduced phosphorylation of protein kinase B (pAKT). This protein is involved in suppression of intracellular lipolysis and NEFA release. Sleep restriction can also alter whole body substrate metabolism such that there is a trend for increased lipid oxidation. Additionally, research examining the effects of short-term sleep restriction on circulating lipids have had mixed results. A number of studies have found decreases in fasting TG while other studies found no change in plasma TGs with sleep restriction.

Aerobic exercise has beneficial effects on postprandial lipemia and insulinemia in normal-weight and obese individuals. Acute moderate-intensity aerobic exercise (30-90 min) performed 12-18 h before an oral fat tolerance test or mixed meal test reduces postprandial TG and insulin concentrations. This response is largely dependent upon the exercise-induced energy deficit as the response is abolished when the calories expended during exercise are replaced.

However, it is not known if sleep restriction will interfere with the beneficial effects of prior exercise on postprandial lipemia. The aim of this project is to investigate if sleep restriction negates the positive effect that exercise has on postprandial lipemia. It is hypothesized that sleep restriction will negate the beneficial effects of prior exercise on postprandial lipemia. Additionally sleep restriction will result in a worsening of the lipid profile compared to no exercise.

For the proposed study, the investigators will use a repeated measures ANOVA (4 study conditions (no exercise+ sleep restriction, no exercise+normal sleep, exercise+normal sleep, exercise+sleep restriction) x time will be used to analyze changes in NEFA and triglyceride (TG) concentrations while a one way ANOVA will be used to analyze area under the curve of the NEFA and TG concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese men and women
* 21-45 years of age
* BMI of 25-35 kg/m2
* Normal sleeping habits of 7-9 hours per night

Exclusion Criteria:

* type 2 diabetic
* diagnosed with cardiovascular disease
* hypertensive
* smokers
* pregnant
* taking lipid-lowering medications
* sleep apnea
* fragmented sleep
* have any recent changes in hormonal birth control
* night shift workers or take regular daytime naps
* any medications known to impact metabolism, appetite, or sleep
* any allergies to milk, ice cream, peanut butter and soy.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
area under the curve of fatty acids concentrations | 4 hour
  blood samples for free fatty acid concentrations will be taken every 30 minutes for 4 hours
area under the curve of triglycerides concentrations | 4 hour
  blood samples for triglyceride concentrations will be taken every 30 minutes for 4 hours

SECONDARY OUTCOMES:
area under the curve of glucose concentrations | 4 hour
  blood samples for glucose concentrations will be taken every 30 minutes for 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kanaley, PhD, Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - University of Misouri, Columbia, Missouri
  - University of Missouri, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: Yes
We will share deidentifiable data that is collected
Supporting Information: Study Protocol, SAP
Time Frame: The data will not be shared until at least 2 years after data collection is completed. Data will be available for another 3 years

REFERENCES:
- [Derived] Maloney A, McDonald M, Petroski G, Kanaley JA. Effect of sleep restriction, with or without prior evening exercise, on morning postprandial lipemia. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-10. doi: 10.1139/apnm-2024-0535. PMID 40294439